CLINICAL TRIAL: NCT05846412
Title: Catheter Ablation or Percutaneous Mitral Valve Repair to Treat Essential (Moderate/Severe) Functional Mitral Regurgitation in Patients With Atrial Fibrillation - a Pilot Trial
Brief Title: Treatment of Functional Mitral Regurgitation in Patients With Atrial Fibrillation
Acronym: CAMERA-Pilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Prof. Dr. Karl-Heinz Kuck (MD), Principal Investigator, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-2022
Record Dates: First submitted 2023-04-04; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation; Mitral Regurgitation Functional
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhythm Control by Catheter Ablation: (Experimental): Patients randomized to rhythm control with CA will undergo CA of AF.
  Interventions: Other: Catheter Ablation and M-TEER
- M-TEER (Control): (Active Comparator): Patients randomized to the M-TEER group will undergo M-TEER with the MitraClip or PASCAL device to reduce FMR severity.
  Interventions: Other: Catheter Ablation and M-TEER

INTERVENTIONS:
Other: Catheter Ablation and M-TEER — Already included in arm descriptions.

SUMMARY:
The objective of the CAMERA-Pilot trial is to generate a hypothesis for a proper randomized controlled clinical endpoint trial to show the noninferiority of restoration and maintenance of sinus rhythm (via catheter ablation [CA] of AF) vs. mitral transcatheter edge-to-edge repair (M-TEER) in patients with AF and concomitant FMR. Patients will be stratified into ventricular FMR with atrial component and atrial FMR.

DETAILED DESCRIPTION:
Rhythm Control by Catheter Ablation: Patients randomized to rhythm control with CA will undergo CA of AF. The index procedure will comprise pulmonary vein isolation (PVI) using either the cryoballoon or radiofrequency (RF) current or pulsed field ablation at the discretion of the investigator. Additional atrial substrate modification may be performed at the discretion of the investigator.

The objective of rhythm control is to restore sinus rhythm by CA and to maintain sinus rhythm during the 12-month follow-up period. In case of AF recurrence during follow-up, sinus rhythm must be restored as soon as possible, either by adding or changing AADs, electrical cardioversion, or repeat CA.

No attempt will be made to reduce FMR by interventional means. Medical treatment of FMR will follow current guidelines.

M-TEER (Control): Patients randomized to the M-TEER group will undergo M-TEER with the MitraClip or PASCAL device to reduce FMR severity. The intervention will be considered successful if FMR is graded 2+ (moderate) or less by an echocardiography core laboratory in accordance with the 2017 Guidelines of the American Society of Echocardiography and specific guidelines on valvular regurgitation after percutaneous valve repair or replacement.

No attempt will be made to restore sinus rhythm, except for patients who remain symptomatic due to AF during follow-up. Medical treatment of AF will follow current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic ventricular FMR (moderate-to-severe [grade 3+] or severe [4+] by independent echocardiographic core laboratory assessment) due to cardiomyopathy of either ischemic or non-ischemic etiology (LVEF 30-49%), concomitant with AF
* Symptomatic atrial FMR (moderate-to-severe [grade 3+] or severe [4+] by independent echocardiographic core laboratory assessment) due to AF, with normal (≥50%) LVEF
* LV end-systolic diameter ≤70 mm
* Documented history of paroxysmal AF (PAF) or persistent AF for maximally 2 years
* Subject has been adequately treated medically for at least 4 weeks per applicable standards, including for coronary artery disease, LV dysfunction, mitral regurgitation and heart failure
* NYHA functional class II, III or ambulatory IV
* Local heart team has determined that MV surgery is not indicated as a treatment option or will be high risk
* Age 18-80 years

Exclusion Criteria:

* Untreated clinically significant coronary artery disease requiring revascularization
* CABG, PCI or TAVR within prior 30 days
* Aortic or tricuspid valve disease (tricuspid regurgitation ≥3+) requiring surgery or transcatheter intervention
* Cerebrovascular accident within prior 30 days
* Severe symptomatic carotid stenosis (>70% by ultrasound)
* Carotid surgery or stenting within prior 30 days
* NYHA functional class IV requiring in-hospital care
* Implant of CRT or CRT-D within the last 30 days
* Transseptal puncture anatomically not feasible
* Leaflet anatomy which may preclude MitraClip/PASCAL implantation, proper MitraClip/PASCAL positioning on the leaflets, or sufficient reduction in mitral regurgitation by the MitraClip/PASCAL device.
* Current pregnancy or planned pregnancy within next 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
FMR grade ≤2+ (moderate or less) at 1 year | 24 Month
  The FMR grade will be assessed with transesophageal echocardiography